CLINICAL TRIAL: NCT01182792
Title: Chronic Hypoxemia and Systemic Vascular Function
Brief Title: Chronic Mountain Sickness, Systemic Vascular Function
Acronym: CMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: Instituto Boliviano de Biologia de Altura (Unknown); Universitad Major de S. Andres, La Paz, Bolivia (Unknown)
Responsible Party: Principal Investigator, Urs Scherrer, Prof, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMS
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Mountain Sickness; Chronic
Keywords: Endothelial Function; Chronic Hypoxia; Oxidative Stress
MeSH Terms: conditions — Altitude Sickness; Bronchiolitis Obliterans Syndrome | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Antioxidant (Experimental)
  Interventions: Dietary Supplement: Vitamin C and E
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C and E — 1 month, 1g Vitamin C and 400 IE Vitamin E or Acute, 1g Vitamin C (in the offspring)
  Arms: Antioxidant
Dietary Supplement: Placebo — 1 month Placebo
  Arms: Control

SUMMARY:
Diseases associated with chronic hypoxemia like chronic obstructive pulmonary disease (COPD) or emphysema, represent major medical and socio-economical problems and one of the leading cause of morbidity and mortality in the western countries. Recently, is has been shown that cardiovascular (CV) diseases contribute highly to the morbidity and mortality of these patients. Furthermore, increasing evidence suggest that systemic vascular dysfunction play a central role in the mediation of the increased CV risk in patients with COPD. However the underlying mechanisms of vascular dysfunction in these patients are incompletely understood. Chronic mountain sickness (CMS) is characterized by chronic hypoxemia related at least in part to hypoventilation; it affects relatively young adults, and may therefore allow to study the effects of chronic hypoxemia. The investigators therefore will assess systemic vascular function and test the hypothesis that increased oxidative stress is responsible for this dysfunction. Since polyglobulia is a hallmark of chronic hypoxemia and has been suggested to affect vascular function, the investigators will test the effects of hemodilution on vascular function. Then, the investigators will test the effects of acute oxygen application and 1 month antioxidative dietary supplement on vascular function.

Preliminary data suggest that offspring of CMS patients may display pulmonary and systemic vascular dysfunction. Antioxidant administration is know to improve vascular function. We will test the acute effect of Vitamin C in this setting.

Finally, since there is considerable inter-individual variability of pulmonary artery pressure among CMS patients and the presence of a patent foramen ovale (PFO)is increased in clinical conditions associated with pulmonary hypertension and hypoxemia, we will assess the prevalence of PFO in healthy high altitude dwellers and in CMS patients and its effects on pulmonary artery pressure at rest and during mild exercise.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Mountain Sickness and their offspring

Exclusion Criteria:

* Smoking
* Lung disease
* Arterial Hypertension

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-10; Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Endothelial Function | 1 month

CONTACTS AND LOCATIONS:
Locations (2):
- Istituto Boliviano de Biologia de Altura, Universitad S. Andres, La Paz, Bolivia
- University Hospital Lausanne, Botnar Center for Extreme Medicine, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Bailey DM, Culcasi M, Filipponi T, Brugniaux JV, Stacey BS, Marley CJ, Soria R, Rimoldi SF, Cerny D, Rexhaj E, Pratali L, Salmon CS, Jauregui CM, Villena M, Villafuerte F, Rockenbauer A, Pietri S, Scherrer U, Sartori C. EPR spectroscopic evidence of iron-catalysed free radical formation in chronic mountain sickness: Dietary causes and vascular consequences. Free Radic Biol Med. 2022 May 1;184:99-113. doi: 10.1016/j.freeradbiomed.2022.03.028. Epub 2022 Apr 6. PMID 35398201
- [Derived] Rexhaj E, Rimoldi SF, Pratali L, Brenner R, Andries D, Soria R, Salinas C, Villena M, Romero C, Allemann Y, Lovis A, Heinzer R, Sartori C, Scherrer U. Sleep-Disordered Breathing and Vascular Function in Patients With Chronic Mountain Sickness and Healthy High-Altitude Dwellers. Chest. 2016 Apr;149(4):991-8. doi: 10.1378/chest.15-1450. Epub 2016 Jan 12. PMID 26540612
- [Derived] Brenner R, Pratali L, Rimoldi SF, Murillo Jauregui CX, Soria R, Rexhaj E, Salinas Salmon C, Villena M, Romero C, Sartori C, Allemann Y, Scherrer U. Exaggerated pulmonary hypertension and right ventricular dysfunction in high-altitude dwellers with patent foramen ovale. Chest. 2015 Apr;147(4):1072-1079. doi: 10.1378/chest.14-1353. PMID 25375664
- [Derived] Pratali L, Allemann Y, Rimoldi SF, Faita F, Hutter D, Rexhaj E, Brenner R, Bailey DM, Sartori C, Salmon CS, Villena M, Scherrer U, Picano E, Sicari R. RV contractility and exercise-induced pulmonary hypertension in chronic mountain sickness: a stress echocardiographic and tissue Doppler imaging study. JACC Cardiovasc Imaging. 2013 Dec;6(12):1287-97. doi: 10.1016/j.jcmg.2013.08.007. Epub 2013 Oct 23. PMID 24269266
- [Derived] Bailey DM, Rimoldi SF, Rexhaj E, Pratali L, Salinas Salmon C, Villena M, McEneny J, Young IS, Nicod P, Allemann Y, Scherrer U, Sartori C. Oxidative-nitrosative stress and systemic vascular function in highlanders with and without exaggerated hypoxemia. Chest. 2013 Feb 1;143(2):444-451. doi: 10.1378/chest.12-0728. PMID 22922469
- [Derived] Pratali L, Rimoldi SF, Rexhaj E, Hutter D, Faita F, Salmon CS, Villena M, Sicari R, Picano E, Allemann Y, Scherrer U, Sartori C. Exercise induces rapid interstitial lung water accumulation in patients with chronic mountain sickness. Chest. 2012 Apr;141(4):953-958. doi: 10.1378/chest.11-0084. Epub 2011 Sep 1. PMID 21885723
- [Derived] Rimoldi SF, Rexhaj E, Pratali L, Bailey DM, Hutter D, Faita F, Salinas Salmon C, Villena M, Nicod P, Allemann Y, Scherrer U, Sartori C. Systemic vascular dysfunction in patients with chronic mountain sickness. Chest. 2012 Jan;141(1):139-146. doi: 10.1378/chest.11-0342. Epub 2011 Jun 23. PMID 21700688